CLINICAL TRIAL: NCT05793515
Title: "Understanding Genetic Missing Variability and Pathogenetic Mechanisms of Inherited Retinal Dystrophies Using Whole Genome Sequencing and in Vitro and in Vivo Models"
Brief Title: Mechanisms of Inherited Retinal Dystrophies Using Whole Genome Sequencing and in Vitro and in Vivo Models
Status: Completed | Type: Observational
Sponsor: Istituto Superiore di Sanità (Other)
Collaborators: Fondazione G.B. Bietti, IRCCS (Other); Ospedale Pediatrico Bambin Gesù (Other)
Responsible Party: Principal Investigator, Viviana Cordeddu, PhD, Istituto Superiore di Sanità
Other Study IDs: ISS20-5656c541c257
Record Dates: First submitted 2023-03-20; First posted 2023-03-31 (Actual); Last update posted 2025-04-18 (Actual); Status verified 2025-04

CONDITIONS: Inherited Retinal Dystrophy; Retinitis Pigmentosa; Macular Dystrophy
Keywords: IRD, RP, WGS, molecular diagnosis
MeSH Terms: conditions — Retinitis Pigmentosa; Macular Degeneration

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples, saliva samples
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (30):
- FB_001: Proband affected by IRD and affected and/or unaffected relatives without molecular diagnosis.
  Interventions: Diagnostic Test: whole genome sequencing
- FB_002: Proband affected by IRD and affected and/or unaffected relatives without molecular diagnosis.
  Interventions: Diagnostic Test: whole genome sequencing
- FB_003: Proband affected by IRD and affected and/or unaffected relatives without molecular diagnosis.
  Interventions: Diagnostic Test: whole genome sequencing
- FB_004: Proband affected by IRD and affected and/or unaffected relatives without molecular diagnosis.
  Interventions: Diagnostic Test: whole genome sequencing
- FB_005: Proband affected by IRD and affected and/or unaffected relatives without molecular diagnosis.
  Interventions: Diagnostic Test: whole genome sequencing
- FB_006: Proband affected by IRD and affected and/or unaffected relatives without molecular diagnosis.
  Interventions: Diagnostic Test: whole genome sequencing
- FB_007: Proband affected by IRD and affected and/or unaffected relatives without molecular diagnosis.
  Interventions: Diagnostic Test: whole genome sequencing
- FB_008: Proband affected by IRD and affected and/or unaffected relatives without molecular diagnosis.
  Interventions: Diagnostic Test: whole genome sequencing
- FB_009: Proband affected by IRD and affected and/or unaffected relatives without molecular diagnosis.
  Interventions: Diagnostic Test: whole genome sequencing
- FB_0010: Proband affected by IRD and affected and/or unaffected relatives without molecular diagnosis.
  Interventions: Diagnostic Test: whole genome sequencing
- FB_0011: Proband affected by IRD and affected and/or unaffected relatives without molecular diagnosis.
  Interventions: Diagnostic Test: whole genome sequencing
- FB_0012: Proband affected by IRD and affected and/or unaffected relatives without molecular diagnosis.
  Interventions: Diagnostic Test: whole genome sequencing
- FB_0013: Proband affected by IRD and affected and/or unaffected relatives without molecular diagnosis.
  Interventions: Diagnostic Test: whole genome sequencing
- FB_0014: Proband affected by IRD and affected and/or unaffected relatives without molecular diagnosis.
  Interventions: Diagnostic Test: whole genome sequencing
- FB_0015: Proband affected by IRD and affected and/or unaffected relatives without molecular diagnosis.
  Interventions: Diagnostic Test: whole genome sequencing
- FB_0016: Proband affected by IRD and affected and/or unaffected relatives without molecular diagnosis.
  Interventions: Diagnostic Test: whole genome sequencing
- FB_0017: Proband affected by IRD and affected and/or unaffected relatives without molecular diagnosis.
  Interventions: Diagnostic Test: whole genome sequencing
- FB_0018: Proband affected by IRD and affected and/or unaffected relatives without molecular diagnosis.
  Interventions: Diagnostic Test: whole genome sequencing
- FB_0019: Proband affected by IRD and affected and/or unaffected relatives without molecular diagnosis.
  Interventions: Diagnostic Test: whole genome sequencing
- FB_0020: Proband affected by IRD and affected and/or unaffected relatives without molecular diagnosis.
  Interventions: Diagnostic Test: whole genome sequencing
- FB_0021: Proband affected by IRD and affected and/or unaffected relatives without molecular diagnosis.
  Interventions: Diagnostic Test: whole genome sequencing
- FB_0022: Proband affected by IRD and affected and/or unaffected relatives without molecular diagnosis.
  Interventions: Diagnostic Test: whole genome sequencing
- FB_0023: Proband affected by IRD and affected and/or unaffected relatives without molecular diagnosis.
  Interventions: Diagnostic Test: whole genome sequencing
- FB_0024: Proband affected by IRD and affected and/or unaffected relatives without molecular diagnosis.
  Interventions: Diagnostic Test: whole genome sequencing
- FB_0025: Proband affected by IRD and affected and/or unaffected relatives without molecular diagnosis.
  Interventions: Diagnostic Test: whole genome sequencing
- FB_0026: Proband affected by IRD and affected and/or unaffected relatives without molecular diagnosis.
  Interventions: Diagnostic Test: whole genome sequencing
- FB_0027: Proband affected by IRD and affected and/or unaffected relatives without molecular diagnosis.
  Interventions: Diagnostic Test: whole genome sequencing
- FB_0028: Proband affected by IRD and affected and/or unaffected relatives without molecular diagnosis.
  Interventions: Diagnostic Test: whole genome sequencing
- FB_0029: Proband affected by IRD and affected and/or unaffected relatives without molecular diagnosis.
  Interventions: Diagnostic Test: whole genome sequencing
- FB_0030: Proband affected by IRD and affected and/or unaffected relatives without molecular diagnosis.
  Interventions: Diagnostic Test: whole genome sequencing

INTERVENTIONS:
Diagnostic Test: whole genome sequencing — Whole genome sequencing will be performed in patients whose test was negative for the targeted resequencing and/or clinical exome sequencing.

SUMMARY:
Inherited retinal dystrophies (IRDs), a large group of heterogeneous and rare disorders, may result in irreversible bilateral visual loss and blindness. Characterizing the genetic bases of IRDs will help to understand the pathogenesis underlying the development of retinal damage. Despite the advances in molecular identification of genes causing disease, unsolved IRDs constitute about 40% of all cases.

Goal of this study is to solve missing heritability in IRD using whole genome sequencing (WGS) to identify the genetic causes in clinically well-characterized patients without a molecular diagnosis.

The identiﬁcation of novel genes that have a role in the development or maintenance of retinal function will lead to the development of new therapeutic approaches and will favour a more prompt diagnosis and improvement of patient management.

DETAILED DESCRIPTION:
IRDs are rare neurodegenerative and genetically heterogeneous conditions with a wide spectrum of presentations, even among affected members of the same family. These disorders exhibit a large range of phenotypes with signiﬁcant overlap, that can be broadly divided into three main groups: those principally affecting the periphery such as retinitis pigmentosa (RP) and choroideremia; those primarily involving the macula, known as 'macular' or 'central' dystrophies; and those affecting both the centre and periphery as seen in cone-rod or rod-cone dystrophies. Collectively, IRDs have an incidence of 1:2000, impacting approx. 2 million people worldwide and patients are progressively visually impaired. Affected individuals can be followed-up by visual acuity measurements, visual field evaluations, electroretinography recordings (ERG), structural imaging with autofluorescence, spectral-domain optical coherence tomography (OCT), and OCT angiography. Although an accurate clinical diagnosis can be reached by these innovative and non-invasive tools, genetic testing is necessary to confirm a specific phenotype, and segregation analysis can address the inheritance pattern. Gene discovery approaches clarified that mutations of about 280 different genes involved in eyes development, photoreceptor survival, phototransduction mechanisms, retinoid cycle, retinal enzymatic function, or cell structure are responsible for these degenerative diseases (RetNet. Available at: https://sph.uth.edu/retnet/) and the inheritance pattern can be autosomal dominant, recessive, or X-linked.

To improve the success rate of genetic/genomic diagnosis, new sequencing technologies have been explored, starting from targeted sequencing focused on multigene panels to whole exome sequencing (WES) and sequencing of the entire genome (WGS). Because of the genetic heterogeneity of IRDs, the congruence of clinical and molecular diagnosis is a necessary goal to characterize exactly the phenotype and to increase the chance of therapeutically beneficial strategies.

A major challenge consists in identifying novel genes encoding for the diseases. This extreme genetic heterogeneity accounts for about 30% of the detection failure of molecular diagnosis. With the possibility of investigating WES or WGS, broader windows are opened for gene discovery.

ELIGIBILITY:
Inclusion Criteria:

* Patients with retinal and optic nerve dystrophy of suspected hereditary nature.
* Probands with clinical follow-up of at least 12 months.
* Patients with an inconclusive molecular diagnosis by means of molecular-genetic tests for the genes known to date for the diagnosed pathology.

Exclusion Criteria:

* Patients with a clinical diagnosis of no proven genetic origin.
* Patients whose parents' or second degree relatives' samples are not available.
* Patients who refuse to be informed of the genetic results obtained, including incidental clinically relevant, validated and actionable for the patient himself and/or his family.

Ages: 5 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Male and female patients, aged between 5 and 80 years, suffering from retinal or optic nerve degeneration of a hereditary nature. Patients will be recruited at the IRCSS Fondazione Bietti in Rome and undergo ophthalmological examinations and instrumental tests. Candidate subjects are a clinically well-characterized cohort of patients with ocular dystrophies, including IRDs already clinically followed for at least 12 months and without a conclusive molecular diagnosis.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2022-11-15 (Actual); Primary Completion 2024-11-02 (Actual); Study Completion 2024-11-02 (Actual)

PRIMARY OUTCOMES:
Understanding genetic missing pathogenetic variants in IRD | two years
  Identification of genetic variants causative of the clinical phenotype

SECONDARY OUTCOMES:
Gene discovery in IRD | two years
  Identification of novel disease genes responsible for IRD.

OTHER OUTCOMES:
Assessment of the pathogenicity of the newly identified variant(s) by functional studies. | three years
  Functional characterization of new variants by in vivo and in vitro models

CONTACTS AND LOCATIONS:
Overall Officials: Viviana Cordeddu, PhD, Principal Investigator — Istituto Superiore di Sanità
Locations (1):
- Istituto Superiore di Sanità-Dpt. Oncology and Molecular Medicine, Rome, Italy, Italy

IPD SHARING:
Plan to Share IPD: Undecided
We plan to share anonymized genomic data among the three partners involved in the study by telecall meetings and shared cloud folders.

REFERENCES:
- [Derived] Brugger M, Lauri A, Zhen Y, Gramegna LL, Zott B, Sekulic N, Fasano G, Kopajtich R, Cordeddu V, Radio FC, Mancini C, Pizzi S, Paradisi G, Zanni G, Vasco G, Carrozzo R, Palombo F, Tonon C, Lodi R, La Morgia C, Arelin M, Blechschmidt C, Finck T, Sorensen V, Kreiser K, Strobl-Wildemann G, Daum H, Michaelson-Cohen R, Ziccardi L, Zampino G, Prokisch H, Abou Jamra R, Fiorini C, Arzberger T, Winkelmann J, Caporali L, Carelli V, Stenmark H, Tartaglia M, Wagner M. Bi-allelic variants in SNF8 cause a disease spectrum ranging from severe developmental and epileptic encephalopathy to syndromic optic atrophy. Am J Hum Genet. 2024 Mar 7;111(3):594-613. doi: 10.1016/j.ajhg.2024.02.005. Epub 2024 Feb 28. PMID 38423010